CLINICAL TRIAL: NCT02898350
Title: Multi-Center Study to Compare the Safety and Efficacy of Clearance of Surgical Scars With the Pulse Dye Laser in Combination With a CO2 Laser in a Split Scar Evaluation
Brief Title: Surgical Scar Treatment With the Pulsed Dye Laser in Combination With a CO2 Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DHF05911
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Scars
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pulsed Dye Laser treatment (Active Comparator): Pulsed Dye Laser treatment after suture removal (3 sessions)
  Interventions: Device: Pulsed dye laser treatment
- CO2 laser treatment (Active Comparator): CO2 laser (3 treatment sessions) after suture removal
  Interventions: Device: CO2 laser treatment
- Combined PDL and CO2 Laser treatment (Active Comparator): Combined PDL and CO2 Laser resurfacing (3 treatment sessions) after suture removal
  Interventions: Device: Combined PDL and CO2 laser treatment
- Split PDL and CO2 Laser treatment (Active Comparator): Half of the scar was not treated and served as a control, while the other half was treated with CO2 ablative fractional resurfacing immediately after surgery, in addition to the three combined PDL and CO2 treatment sessions after suture removal
  Interventions: Device: Split PDL and CO2 Laser treatment

INTERVENTIONS:
Device: Pulsed dye laser treatment — Scar minimization with Pulsed dye laser treatment on suture removal day
  Other Names: Vbeam, Vbeam Perfecta, PDL
  Arms: Pulsed Dye Laser treatment
Device: CO2 laser treatment — Scar minimization with CO2 laser treatment on suture removal day
  Other Names: CO2RE, CORE
  Arms: CO2 laser treatment
Device: Combined PDL and CO2 laser treatment — Scar minimization with Pulsed dye laser and CO2 laser treatment on suture removal day
  Other Names: Vbeam, Vbeam Perfecta, CO2RE, CORE
  Arms: Combined PDL and CO2 Laser treatment
Device: Split PDL and CO2 Laser treatment — Split-scar with CO2 treatment after surgery and combined PDL and CO2 treatment on suture removal day
  Arms: Split PDL and CO2 Laser treatment

SUMMARY:
Prospective, randomized, split lesion treatment with 4 study Arms to evaluate safety and efficacy of combined treatment for minimizing of surgical scars, including post Moh's surgery.

DETAILED DESCRIPTION:
Prospective, Randomized, Split lesion treatment with 4 study Arms: 1) treatment with pulsed dye laser (PDL) only, 2) treatment with CO2 laser only, 3) PDL and CO2 laser combined treatment, and 4) split scar combined lasers with an additional single CO2 laser treatment immediately post-surgery vs. no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Comprehension of, and willingness to sign, the Informed Consent Form.
* Have a planned a surgical procedure, which is expected to result in a least one linear surgical scar of at least 3.0 cm.
* Be a healthy male or female of at least 18 years old.
* Fitzpatrick skin type I-V.
* Willingness to follow the treatment and follow-up schedule and the post-treatment care instructions.
* Non pregnant and/or breast feeding, if applicable.
* Willingness to provide a brief medical history including disclosure of any prescribed or over-the-counter medications taken within the past 6 months.
* Agree to follow and undergo all study-related procedures.
* Use of daily use of sunblock SPF 30 or higher for duration of the study.

Exclusion Criteria:

1. Pregnant and/or breastfeeding.
2. Fitzpatrick skin type VI.
3. Prior treatment for the surgical scar to be treated in this study.
4. Having a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen.
5. Use of Isotretinoin or other systemic retinoids within the past 6 months.
6. Use of topical retinoids or therapeutic topicals in the treatment area in past 2 months.
7. Use of medications that induce photosensitivity on the 595 and 10,600 nm wavelength ranges.
8. Suffering from current or history of significant skin conditions in the treated area or inflammatory skin conditions.
9. History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
10. Having any uncontrolled disease or disorder or one which per the investigator's judgment might make it unsafe for the subject to participate in this study.
11. Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning and sun exposure for the duration of the study.
12. Participation in another investigational device or investigational drug study within 30 days prior to enrollment, as per the investigator's clinical judgment.
13. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-02; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Improvement in Global Evaluation Response (GER) scale for 4 study arms compared to baseline | Baseline, 3 months after final treatment
  Blinded review of 7-point Global Evaluation Response (GER) scale

SECONDARY OUTCOMES:
Improvement in Vancouver Scar Scale (VSS) scale for 4 study arms compared to baseline | Baseline, 3 months after final treatment
  Investigator review of VSS - The VSS assesses four variables: vascularity, pigmentation, pliability, and height of the scar, to provide an overall score from 0 (normal) to 13 (severe).

OTHER OUTCOMES:
Number and severity of adverse events | Baseline and up to 3 months after treatment
  Number and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Shlomit Mann, MSc, Study Director — Syneron Medical
Locations (2):
- United States (2):
  - AboutSkin, Dermatology and Derm Surgery PC, Englewood, Colorado
  - Laser & Skin Surgery Center of New York, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cohen JL. Minimizing skin cancer surgical scars using ablative fractional Er:YAG laser treatment. J Drugs Dermatol. 2013 Oct;12(10):1171-3. PMID 24085055
- [Background] Weiss ET, Chapas A, Brightman L, Hunzeker C, Hale EK, Karen JK, Bernstein L, Geronemus RG. Successful treatment of atrophic postoperative and traumatic scarring with carbon dioxide ablative fractional resurfacing: quantitative volumetric scar improvement. Arch Dermatol. 2010 Feb;146(2):133-40. doi: 10.1001/archdermatol.2009.358. PMID 20157023
- [Background] Alster T. Laser scar revision: comparison study of 585-nm pulsed dye laser with and without intralesional corticosteroids. Dermatol Surg. 2003 Jan;29(1):25-9. doi: 10.1046/j.1524-4725.2003.29024.x. PMID 12534508